CLINICAL TRIAL: NCT05515315
Title: Induction Tislelizumab Combined With Chemotherapy Followed by Definitive Chemoradiotherapy in the Treatment of Locally Unresectable Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPT-ESCC
Record Dates: First submitted 2022-08-19; First posted 2022-08-25 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Immunotherapy Esophagus Cancer
MeSH Terms: interventions — tislelizumab; nedaplatin; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab combined with chemothapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Albumin paclitaxel; Drug: Nedaplatin; Radiation: radiotherapy

INTERVENTIONS:
Drug: Tislelizumab — Participants will receive Tislelizumab, 200mg, intravenously over 30 - 60 minutes, day 1 of every 3 weeks
Drug: Albumin paclitaxel — Participants will receive Albumin paclitaxel 260 mg/m2 , day 1 of every 3 weeks
Drug: Nedaplatin — Participants will receive Nedaplatin 80 mg/m2 , day 1 of every 3 weeks
Radiation: radiotherapy — 50-60Gy/25-30f

SUMMARY:
To explore the efficacy of Tislelizumab combined with chemotherapy in the treatment of locally unresectable esophageal squamous cell carcinoma (ESCC)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed localized ESCC that is suitable for cCRT, including: stage II-IVA (AJCC version 8) inoperable ESCC (medically unfit for surgery or refusing surgical intervention);;
* Aged 18-70, both sexes;
* ECOG score 0-1
* The presence of measurable and/or nonmeasurable lesions that met the definition of RECIST1.1;
* Adequate organ and bone marrow function, meeting the following definitions:

  1. Blood routine (no blood transfusion, no granulocyte colony-stimulating factor [G-CSF], and no other drugs were used within 14 days before treatment);Absolute neutrophil count (ANC) ≥1.5×109/L;Hemoglobin (HB) ≥9.0 g/dL;Platelet count (PLT) ≥100×109/L;
  2. Blood biochemistry Creatinine clearance rate ≥60 mL/min;Total bilirubin (TBIL) ≤ 1.5×ULN;Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤2.5×ULN;
* Expected survival time > 6 months;
* Fertile female subjects and male subjects with partners of reproductive age are required to use a medically approved contraceptive method during the study treatment period and for at least 3 months after the last treatment;
* Patients who volunteered to participate in this study and signed the informed consent form.

Exclusion Criteria:

* A history of fistula caused by primary tumor invasion;
* Presence of clinically uncontrolled pleural effusion, pericardial effusion, or ascites that required repeated drainage or medical intervention (within 2 weeks before randomization);
* Known intolerance or resistance to chemotherapy specified in the trial protocol;
* have received any other ESCC antitumor therapy (e.g., therapy targeting PD-1, PD-L1, PD-L2 or other tumor immunotherapy, radiotherapy, targeted therapy, ablation or other systemic or local antitumor therapy);
* Patients with active autoimmune disease or a history of autoimmune disease that may relapse, or a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* History of interstitial lung disease, non-infectious pneumonia or uncontrolled systemic diseases, including pulmonary fibrosis and acute lung disease;
* Severe chronic or active infection (including tuberculosis infection) requiring systemic antimicrobial therapy, antifungal therapy or antiviral therapy before enrollment;
* Known history of HIV infection;
* Other malignancies (except cured basal cell carcinoma of the skin, carcinoma in situ of the breast and carcinoma in situ of the cervix) in the past 5 years;
* Received live vaccine within 28 days before enrollment;
* while participating in another therapeutic clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
progression free survival | up to 24 months
  Time from enrollment to the onset of disease progression or death

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | every 6 weeks （up to 24 months）
  Objective Response Rate Determine the tumor shrinkage rate, tumor boundary and the adhesion of tumor
Overall survival (OS) | every 3 months (up to 24 months)
  Defined from date of Signing ICF to date of first documentation of death from any cause or censored at the date of the last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Ye zai sheng, Fuzhou, Fujian, China